CLINICAL TRIAL: NCT03201861
Title: Phase 3 Study of Weekly Paclitaxel in Combination With Cisplatin as Adjuvant Chemotherapy for Early Stage Human Epidermal Growth Factor Receptor-2 (HER2) Negative Breast Cancer in High-risk Women
Brief Title: Addition of Cisplatin to Adjuvant Chemotherapy for Early Stage Breast Cancer in High-Risk Women
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHPD004
Record Dates: First submitted 2017-06-08; First posted 2017-06-28 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Tubular Breast Cancer; Mucinous Breast Cancer; Invasive Duct Carcinoma of Breast
MeSH Terms: conditions — Carcinoma, Ductal, Breast | interventions — TP protocol; Paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- paclitaxel and cisplatin (Experimental): Drug: paclitaxel, cisplatin, epirubicin and cyclophosphamide Patients will be administered paclitaxel (80 mg/m² i.v. given weekly on day 1 q day 8 for 12 weeks) and cisplatin (25 mg/m² weekly on day 1 ,8,and 15 q day 28 for 3 cycles) followed by epirubicin and cyclophosphamide (EC) (epirubicin 90mg/m² i.v.d1, cyclophosphamide 600mg/m² i.v.d1) for 4 cycles.
  Interventions: Drug: Paclitaxel, Cisplatin
- epirubicin and cyclophosphamide (Active Comparator): Drug：epirubicin, cyclophosphamide, paclitaxel and docetaxel
  Investigators will declare one of the following regimens:
  Patients with hormone receptor (HR) positive breast cancer wil be administered epirubicin (90mg/m² i.v.d1 q21d) and cyclophosphamide (600mg/m² i.v.d1 q21d) for 4 cycles followed by docetaxel (75mg/m² i.v.d1 q21d) for 4 cycles.
  Patients with triple-negative breast cancer will be administered epirubicin (90mg/m² i.v.d1 q21d) and cyclophosphamide (600mg/m² i.v.d1 q21d) for 4 cycles followed by weekly paclitaxel (80 mg/m² i.v.d1) for 12 weeks or docetaxel (75mg/m² i.v.d1 q21d) for 4 cycles.
  Interventions: Drug: EC to docetaxel or paclitaxel

INTERVENTIONS:
Drug: Paclitaxel, Cisplatin — weekly paclitaxel and cisplatin
  Other Names: Taxol
  Arms: paclitaxel and cisplatin
Drug: EC to docetaxel or paclitaxel — Standard adjuvant chemotherapy recommended by guideline
  Other Names: Taxol
  Arms: epirubicin and cyclophosphamide

SUMMARY:
The investigators hypotheses that paclitaxel combined with cisplatin in a weekly-based regimen as adjuvant chemotherapy is more effective for high risk, HER2 negative breast cancer .

DETAILED DESCRIPTION:
In this trial, patients will be randomly assigned in a 2:1 ratio to receive cisplatin-based adjuvant chemotherapy and to standard adjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged ≥18 years and ≤70 years
2. Have accepted surgical treatment, histologically confirmed early breast cancer, the pathological types of invasive carcinoma
3. Not received treatment for breast cancer before operation
4. Triple-negative breast cancer confirmed by pathology, or pathology confirmed as the HR positive breast cancer at the same time meet the following conditions: axillary lymph node positive breast cancer, tumor size≥2 cm and Ki - 67 >20% or tumor size ≥2 cm and grade III or tumor size ≥2cm and aged <35 years
5. HER2 negative: immunohistochemistry HER2 (1 +) or HER2 (0), or fluorescence in situ hybridization (FISH): not amplified
6. Performance status (PS) 0-1
7. Adequate bone marrow function:WBC≥4.0×109/L, Absolute neutrophil count（ANC）≥1.5×109/L, Platelets（PLT）≥100×109/L, Hemoglobin（Hb）≥90g/L;aspartate aminotransferase(AST),Alanine aminotransferase (ALT)≤1.5 upper normal limit , creatinine≤1.5 upper normal limit, bilirubin≤1.5 upper normal limit
8. No obvious main organs dysfunction

Exclusion Criteria:

1. metastatic breast cancer
2. Patient is pregnant or breast feeding
3. Any evidence of sense or motor nerve disorders
4. Bilateral Primary Breast Cancer (DCIS in one side not included)
5. Patients with medical conditions taht indicate intolerant to adjuvant chemotherapy, including uncontrolled cardiovascular disease, severe infection
6. Have received chemotherapy because of any malignancy other than breast cancer
7. Known severe hypersensitivity to any drugs in this study

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 762 (Estimated)
Dates: Start 2017-07-27 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Disease-Free Survival (DFS) Events | up to 5 year follow up
  DFS is defined as the time period between registration and first event

SECONDARY OUTCOMES:
Number of Participants With Overall Survival (OS) Events | up to 5 year follow up
  OS is defined as the time period between registration and first event
Number of participants with treatment-related adverse events as assessed by CTCAE v3.0. | 5 months during adjuvant therapy
  Descriptive statistics for the treatment will be given on the number of patients whose treatment had to be reduced, delayed or permanently stopped

CONTACTS AND LOCATIONS:
Overall Officials: Jinsong Lu, M.D., Principal Investigator — Shanghai Jiao Tong University School of Medicine
Locations (1):
- Renji Hospital, School of Medicine, Shanghai Jiaotong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sparano JA, Zhao F, Martino S, Ligibel JA, Perez EA, Saphner T, Wolff AC, Sledge GW Jr, Wood WC, Davidson NE. Long-Term Follow-Up of the E1199 Phase III Trial Evaluating the Role of Taxane and Schedule in Operable Breast Cancer. J Clin Oncol. 2015 Jul 20;33(21):2353-60. doi: 10.1200/JCO.2015.60.9271. Epub 2015 Jun 15. PMID 26077235